CLINICAL TRIAL: NCT04258761
Title: A Multi-Center, Open Label, Single Ascending Dose Safety and Tolerability Study of Subcutaneously Administered 10XB-101 in Adult Subjects With Excessive Submental Fat
Brief Title: A Safety and Tolerability Study of 10XB-101 Injections in Adult Subjects With Extra Fat Under the Chin ("Double Chin")
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 10xBio, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 210-9451-202
Record Dates: First submitted 2020-01-27; First posted 2020-02-06 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Submental Fat
MeSH Terms: interventions — Injections; Polidocanol

STUDY DESIGN:
Intervention Model Description: Multi-center, open label, single ascending dose comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 10XB-101 Solution for Injection 1.25% (Experimental): Participants receive 10XB-101 Solution for Injection, 1.25% via subcutaneous injection up to 10 mL on Day 1 of subject participation.
  Interventions: Drug: 10XB-101 Solution for Injection
- 10XB-101 Solution for Injection 2.0% (Experimental): Participants receive 10XB-101 Solution for Injection, 2.0% via subcutaneous injection up to 10 mL on Day 1 of subject participation.
  Interventions: Drug: 10XB-101 Solution for Injection
- 10XB-101 Solution for Injection 3.0% (Experimental): Participants receive 10XB-101 Solution for Injection, 3.0% via subcutaneous injection up to 10 mL on Day 1 of subject participation.
  Interventions: Drug: 10XB-101 Solution for Injection
- 10XB-101 Solution for Injection 4.5% (Experimental): Participants receive 10XB-101 Solution for Injection, 4.5% via subcutaneous injection up to 10 mL on Day 1 of subject participation.
  Interventions: Drug: 10XB-101 Solution for Injection
- 10XB-101 Solution for Injection 6.0% (Experimental): Participants receive 10XB-101 Solution for Injection, 6.0% via subcutaneous injection up to 10 mL on Day 1 of subject participation.
  Interventions: Drug: 10XB-101 Solution for Injection

INTERVENTIONS:
Drug: 10XB-101 Solution for Injection — Active test article
  Other Names: polidocanol

SUMMARY:
The purpose of this research study is to find out more about an investigational drug, 10XB-101, for people with fat under their chin which they would like to remove. The Sponsor of this study thinks there may be a chance this drug could be used to dissolve, or "melt" this fat away.

DETAILED DESCRIPTION:
About 15 subjects with excessive submental fat (SMF) will be enrolled across 2 sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or non-pregnant female 18-65 years of age
* Signed informed consent
* Subject has a score of 2 or 3 on the Clinician Submental Fat Scale (CSFS) at Visit 2/Baseline
* Subject is in good general health

Exclusion Criteria:

* Loose skin or prominent platysmal bands in the neck or chin area
* Recent treatment with anticoagulants
* Presence of clinically significant health problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 24 weeks
  Incidence (severity and causality) of any local and systemic Adverse Events
Local Skin Reactions (LSR) | 24 weeks
  At each time point, the number of subjects with presence (and severity) of the following LSRs on a 4 point scale (zero to 3), with a higher score indicating a worse outcome: erythema, edema, tenderness on palpation, bruising, pain, and stinging/burning

SECONDARY OUTCOMES:
Clinician Submental Fat Scale (CSFS) | 24 weeks
  Change from Baseline in the CSFS on a five-point scale (zero to 4), with a higher score indicating a worse outcome
Patient Submental Fat Scale (PSFS) | 24 weeks
  Change from Baseline in the PSFS on a five-point scale (zero to 4), with a higher score indicating a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: John Dobak, MD, Study Director — 10xBio, LLC
Locations (1):
- Site 01, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No